CLINICAL TRIAL: NCT00656760
Title: The Clinical Utility of PET-CT in the Management of Squamous Cell Carcinoma of Neck Nodes With an Unknown Primary Malignancy.
Brief Title: PET/CT: Role in Detecting Unknown Primary Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Tom Baker Cancer Centre (Other)
Responsible Party: Principal Investigator, Joseph C. Dort, Professor of Surgery, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: UCENT0001
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Head and Neck Cancer
Keywords: unknown primary, head and neck cancer, squamous cell carcinoma; Unknown primary head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): All patients have PET/CT and biopsies with the surgeon blinded to the result of PET/CT. Additional biopsies are performed (or not) after the surgeon has the PET/CT results revealed.
  Interventions: Other: PET/CT

INTERVENTIONS:
Other: PET/CT — PET/CT is being performed on all patients in the study.

SUMMARY:
Historically metastatic squamous cell carcinoma in a cervical lymph node from an occult primary malignancy of the head and neck was evaluated with panendoscopy and biopsies of high risk areas, such as the base of tongue, nasopharynx, and tonsils. This diagnostic protocol identifies the primary malignancy in about 50% of cases. In recent years, the availability of CT has slightly increased the detection rate to 65% when used as an adjunct to the traditional work-up. Studies using PET as an adjunct are conflicting with detection rates ranging up to 75%. Currently, no prospective study has analyzed the role of the PET-CT fusion in the work-up of an occult primary malignancy of the head and neck. This study will compare the detection rate of the traditional work-up to a new protocol involving a pre-operative diagnostic PET-CT.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Biopsy proven SCC in a cervical lymph node
* Unknown primary cancer after: History, Physical exam, and office endoscopy by otolaryngologist
* Negative Chest X-Ray for malignancy
* Patient consent signed to undergo investigative protocol

Exclusion Criteria:

* Un-fit for general anesthesia
* Unable to lie flat for 45 minutes
* Unable to fast for > 6 hours
* Unable to perform PET-CT (Obesity > 150kg)
* Pregnant
* Prior Head and Neck cancer
* Any invasive cancer (Non-Head and Neck) within the last 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
proportion of patients where PET/CT resulted in a change in diagnosis | 2 weeks after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada